CLINICAL TRIAL: NCT01577459
Title: A Phase 1 Crossover Study of Blood Pressure and Heart Rate Response to Pseudoephedrine Concurrent With Placebo or TR 701 FA
Brief Title: A Phase 1 Crossover Study of Blood Pressure and Heart Rate Response
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trius Therapeutics LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 1986-033; TR701-114 (Other: TriusRX Unique ID)
Record Dates: First submitted 2012-04-11; First posted 2012-04-13 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — tedizolid phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TR-701 FA with PSE (Experimental): TR-701 FA 200 mg oral with PSE
  Interventions: Drug: TR-701 FA with PSE
- TR-701 FA Placebo with PSE (Placebo Comparator): TR-701 FA Placebo 200 mg oral with PSE
  Interventions: Other: TR-701 FA Placebo with PSE

INTERVENTIONS:
Drug: TR-701 FA with PSE — TR-701 FA Oral 200 mg oral with PSE
  Other Names: Tedizolid Phosphate
  Arms: TR-701 FA with PSE
Other: TR-701 FA Placebo with PSE — TR-701 FA Placebo Oral 200 mg with PSE
  Arms: TR-701 FA Placebo with PSE

SUMMARY:
This is a randomized, double-blinded, placebo-controlled, crossover study to evaluate the pressor effects of pseudoephedrine when administered with TR-701 FA in healthy adult volunteers.

DETAILED DESCRIPTION:
Eligible subjects will be randomized to 1 of 2 possible treatment sequences (N=9 per sequence) on Study Day 1. Subjects will receive oral 200 mg TR 701 FA or Placebo for TR 701 FA once daily for 5 days during each treatment period, with a 2 day washout between periods (72 hours between doses). On Study Day 5 of each treatment period, subjects will also receive oral 60 mg PSE.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 45 years of age, inclusive
* Healthy males and females with no clinically significant abnormalities identified by a detailed medical history
* Body mass index ≥ 19.0 kg/m2 and ≤ 31.0 kg/m2

Exclusion Criteria:

* Systolic blood pressure > 130 mmHg or < 90 mmHg measured after 10 minutes supine at the Screening Visit and Study Day 1
* Diastolic blood pressure > 90 mmHg or < 60 mmHg measured after 10 minutes supine at the Screening Visit and Study Day 1
* Heart rate > 90 bpm or < 50 bpm measured after 10 minutes supine at the Screening Visit and Study Day
* Known allergy or hypersensitivity to PSE

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-04-23 (Actual); Primary Completion 2012-06-15 (Actual); Study Completion 2012-06-15 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 13 days
  To compare systolic blood pressure post administration of pseudoepherine concurrent with TR-701 FA and Placebo

CONTACTS AND LOCATIONS:
Overall Officials: Philippe G Prokocimer, MD, Study Chair — Trius Therapeutics
Locations (1):
- Trius Investigator Site 001, Overland Park, Kansas, United States

REFERENCES:
- [Result] Flanagan S, Minassian SL, Prokocimer P. Pharmacokinetics of Tedizolid and Pseudoephedrine Administered Alone or in Combination in Healthy Volunteers. J Clin Med. 2018 Jun 14;7(6):150. doi: 10.3390/jcm7060150. PMID 29899212
- [Derived] Flanagan S, Bartizal K, Minassian SL, Fang E, Prokocimer P. In vitro, in vivo, and clinical studies of tedizolid to assess the potential for peripheral or central monoamine oxidase interactions. Antimicrob Agents Chemother. 2013 Jul;57(7):3060-6. doi: 10.1128/AAC.00431-13. Epub 2013 Apr 22. PMID 23612197